CLINICAL TRIAL: NCT00055757
Title: A Phase II Trial of R115777, a Farnesyl Transferase Inhibitor, in Combination With Gemcitabine and Cisplatin in Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Tipifarnib, Gemcitabine, and Cisplatin in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02808; MC0123; N01CM17104 (NIH); N01CM17102 (NIH)
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tipifarnib; Cisplatin; Gemcitabine

ARMS (1):
- Treatment (tipifarnib, gemcitabine, cisplatin) (Experimental): Patients receive oral tipifarnib twice daily on days 1-14, gemcitabine IV over 30 minutes on days 1 and 8, and cisplatin IV over 2 hours on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Patients with at least stable disease may continue to receive oral tipifarnib alone twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tipifarnib; Drug: cisplatin; Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: tipifarnib — Given orally
  Other Names: R115777; Zarnestra
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of combining tipifarnib with gemcitabine and cisplatin in treating patients who have stage III or stage IV non-small cell lung cancer. Drugs used in chemotherapy such as gemcitabine and cisplatin use different ways to stop tumor cells from dividing so they stop growing or die. Tipifarnib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Combining tipifarnib with combination chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the response rate in non-small cell lung cancer (NSCLC) patients receiving combination therapy with R115777, gemcitabine, and cisplatin.

SECONDARY OBJECTIVES:

I. To estimate the time to event efficacy variables including: time to progressive disease, time to treatment failure, time to death of any cause.

II. To estimate the duration of response for responding patients. III. To characterize the toxicities of R115777, gemcitabine, and cisplatin in this patient population.

TERTIARY OBJECTIVES:

I. To evaluate the association between polymorphism expression in candidate genes and clinical endpoints and toxicity to R115777, gemcitabine, and cisplatin.

OUTLINE: This is a multicenter study.

Patients receive oral tipifarnib twice daily on days 1-14, gemcitabine IV over 30 minutes on days 1 and 8, and cisplatin IV over 2 hours on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients with at least stable disease may continue to receive oral tipifarnib alone twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC with one of the following classifications:

  * Stage IIIB with pleural effusion
  * Stage IIIB and not a candidate for combined modality treatment with radiation therapy and chemotherapy
  * Stage IV
* Measurable disease, defined as at least one lesion whose longest diameter can be accurately measured as >= 2.0 cm
* Absolute neutrophil count (ANC) >= 1500/mm^3
* PLT >= 100,000
* Hgb > 10.0 g/dL
* Direct bilirubin =< 1.5 x UNL
* Alkaline phosphatase =< 5 x UNL
* AST =< 3 x UNL
* Creatinine =< 1.5 x UNL
* ECOG Performance Status (PS) 0 or 1
* Capable of understanding the investigational nature, potential risks and benefits of the study and able to provide valid informed consent

Exclusion Criteria:

* Any of the following as this regimen may be harmful to a developing fetus or nursing child:

  * Pregnant women
  * Breastfeeding women
  * Men or women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.)
* Any of the following prior therapies:

  * Prior chemotherapy for NSCLC (exception: therapies used as a radiosensitizer such as low-dose weekly cisplatin and carbo/taxol with XRT)
  * Prior radiation > 25% of bone marrow
  * Prior immunotherapy, biologic or gene therapy
* New York Heart Association classification III or IV
* CNS metastases
* Uncontrolled infection
* Any other severe, underlying diseases that are, in the judgment of the investigator, inappropriate for entry into this study
* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, adequately treated noninvasive carcinomas, or other cancer from which the patient has been disease-free for at least five years
* Pre-existing peripheral neuropathy (motor or sensory) > grade 1 per NCI Common Toxicity Criteria (CTC)
* Known peripheral vascular disease or a history of deep vein thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2003-10; Primary Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Proportion of confirmed tumor responses, defined to be either a CR or PR noted as the objective status on 2 consecutive evaluations at least 4 weeks apart | Up to 18 weeks (6 courses)
  Ninety-five percent confidence intervals for the true success proportion will be calculated.

SECONDARY OUTCOMES:
Survival time | Time from registration to death due to any cause, assessed up to 2 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time to disease progression | Time from registration to documentation of disease progression, assessed up to 2 years
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Duration of response is defined for all evaluable patients who have achieved an objective response as the date at which the patient's objective status is first noted to be either a CR or PR to the date progression is documented | Up to 2 years
Time to treatment failure | Time from the date of registration to the date at which the patient is removed from treatment due to progression, toxicity, or refusal, assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alex Adjei, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States